CLINICAL TRIAL: NCT00003936
Title: Phase II Clinical Evaluation of Bryostatin 1 in Patients With Hodgkin's Disease
Brief Title: Bryostatin 1 in Treating Patients With Recurrent or Refractory Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067128; P30CA022453 (NIH); WSU-C-1902; NCI-T97-0120
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients who have recurrent or refractory Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in patients with recurrent or refractory Hodgkin's disease treated with bryostatin 1. II. Determine qualitative and quantitative toxicities of bryostatin 1 in these patients. III. Determine duration of response and survival in these patients.

OUTLINE: Patients receive bryostatin 1 by continuous IV infusion over 72 hours. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity for at least 4 courses. Patients who achieve complete response (CR) are treated with 4 additional courses beyond CR.

PROJECTED ACCRUAL: A total of 14-27 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of recurrent or refractory Hodgkin's disease Measurable disease Must have failed the following regimens: Mechlorethamine, vincristine, procarbazine, and prednisone (MOPP) AND Doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) May have undergone either bone marrow or peripheral blood stem cell transplant Must not be eligible for standard treatment (high intensity therapy with peripheral blood stem cell or bone marrow transplant) or higher priority protocol

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count (ANC) at least 1,000/mm3 (at least 500/mm3 if extensive bone marrow involvement) Platelets at least 75,000/mm3 (at least 50,000/mm3 if extensive bone marrow involvement) Hepatic: Bilirubin less than 1.5 mg/dL ALT and AST less than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (8 weeks since mitomycin or nitrosoureas) and recovered Endocrine therapy: No concurrent steroids Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Eilender, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States